CLINICAL TRIAL: NCT00675636
Title: Vanderbilt Hereditary Colorectal Cancer Registry
Brief Title: Collecting Information From Patients and Family Members With Hereditary Colorectal Cancer Syndromes or Who Are at High Risk of Developing Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Molly Cone, Assistant Professor, Vanderbilt University Medical Center
Other Study IDs: CDR0000587344; P30CA068485 (NIH); VU-VICC-GI-0721; VU-VICC-061182
Record Dates: First submitted 2008-05-08; First posted 2008-05-09 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-08

CONDITIONS: Colorectal Cancer; Hereditary Non-polyposis Colon Cancer; Precancerous Condition
Keywords: colon cancer; hereditary non-polyposis colon cancer; rectal cancer; familial adenomatous polyposis
MeSH Terms: conditions — Colorectal Neoplasms; Colorectal Neoplasms, Hereditary Nonpolyposis; Precancerous Conditions; Colonic Neoplasms; Rectal Neoplasms; Adenomatous Polyposis Coli

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: study of socioeconomic and demographic variables — database, no intervention
Procedure: evaluation of cancer risk factors — database, no intervention
Procedure: study of high risk factors — database, no intervention

SUMMARY:
RATIONALE: Gathering medical and family history information from patients and family members may help doctors better understand hereditary colorectal cancer and hereditary polyposis syndrome and identify patients at high risk of developing hereditary colorectal cancer.

PURPOSE: This research study is collecting information from patients and family members with hereditary colorectal cancer or polyposis syndrome or who are at high risk of developing hereditary colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To identify patients and their family members who have either hereditary colorectal cancer or polyposis syndrome or are at high risk for developing hereditary colorectal cancer.

Secondary

* To establish a tissue and data repository that will be used to further research in hereditary colorectal cancer syndromes.

OUTLINE: Data is collected on patients and their families for inclusion in a hereditary colorectal cancer registry. Registry data is entered into a secure database that includes information on patient demographics and medical and family cancer history. The information collected will be used to formulate screening and surveillance recommendations, to further knowledge of hereditary colorectal cancer, and to facilitate cancer research. Registry data will also be used to improve the quality of current standard of care through timely tracking and notification of patients for follow-up care, identification of registry participants at high risk for developing an inherited form of colon cancer, and by serving as a resource for future research.

Registry patients may undergo optional blood, urine, and/or sputum sample collection for inclusion in the tissue repository. Tissue samples from a previous biopsy may also be obtained. Samples will be stored for future research studies.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets any of the following criteria:

  * Patients and family members with a known hereditary colorectal cancer or polyposis syndrome
  * Patients who meet Amsterdam I, II, or Bethesda criteria
  * Patients with a family history suggestive of a hereditary colorectal or polyposis syndrome
  * Patients diagnosed with colorectal cancer at < 50 years old
* Patients are identified through surgical, oncological, gynecological, and gastrointestinal programs, as well as outside referrals, self referral, and the Vanderbilit Tumor Registry

PATIENT CHARACTERISTICS:

* See Disease Characteristics

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Anyone with known or suspected hereditary colorectal cancer syndrome, early age o onset of colorectal cancer (see below).
Sampling Method: Non-Probability Sample
Enrollment: 730 (Actual)
Dates: Start 2007-01; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Identification of patients at high risk of developing hereditary colorectal cancer | continuous data collection
  Database will continue indefinitely with IRB approval and investigator support

SECONDARY OUTCOMES:
Establishment of a tissue and data repository | continuous data collection

CONTACTS AND LOCATIONS:
Overall Officials: Paul Wise, MD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee